CLINICAL TRIAL: NCT06736145
Title: Effects of Cervical Nags on Accessory Muscles in Patients With Copd
Brief Title: Cervical Nags Effect on Accessory Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01938 Ghaniya Khan
Record Dates: First submitted 2024-06-12; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: COPD
Keywords: Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Pulmonary Disease; Chronic Obstructive Lung Disease; COPD; COAD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): Cervical stretches and inspiratory muscle training
  Interventions: Other: Traditional Physical Therapy
- Mulligan Glides (Experimental): Mulligan Natural Apophyseal Glides along with cervical stretches and inspiratory muscle training
  Interventions: Other: Mulligan Glides

INTERVENTIONS:
Other: Traditional Physical Therapy — Diaphragmatic, Pursed Lip breathing and Targeted cervical muscle stretches 10 repetitions x 1 set, 3 days/week
  Total of 9 sessions were given each consisting of 40 mins.
  Arms: Traditional Physical Therapy
Other: Mulligan Glides — Natural Apophyseal Glides of Cervical spine are given 3 repetitions x 3-6 sets, 3 days/week.
  Diaphragmatic, Pursed Lip breathing and Targeted cervical muscle stretches 10 repetitions x 1 set, 3 days/week
  Total of 9 sessions were given each consisting of 40 mins.
  Arms: Mulligan Glides

SUMMARY:
The aim of this work is to record changes on accessory muscles especially sternocleidomastoid and scalene after applying cervical NAGs in COPD patients.

DETAILED DESCRIPTION:
Natural gliding movements in the spine, known as apophyseal glides, occur during breathing. These movements are believed to be important for maintaining good posture and flexibility in the spine. In COPD patients, the muscles that support the spine, like the scalene and SCM, can become tight and strained due to labored breathing. This tightness can lead to neck and shoulder pain.

While studies suggest that natural apophyseal glides improve spinal mobility, accessory muscle flexibility and reduce pain, there is room for further research on COPD patients, especially in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Registered with history of moderate (II) to severe (III) grade COPD (for a minimum of 1 year) will be included in the study.
* Patients who are clinically stable.

Exclusion Criteria:

* Patients who have any pre-existing cervical spine disease.
* Patients who have any cardiac disease.
* Other respiratory co-morbidities
* Patients who have severe dizziness or coughing

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Tape Line | 3rd week
  Changes from baseline ROM range of motion for cervical flexion,etension, lateral flexion and rotation is measured using tape
NPRS | 3rd week
  Changes from baseline for pain is measured using NPRS. NPRS stands for Numerical Pain Rating Scale, a common method for assessing pain intensity. It's a simple scale from 0 to 10, where: 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-10 represents severe pain. Patients are asked to rate their pain by choosing a number on this scale to evaluate and monitor pain levels before and after treatment.

SECONDARY OUTCOMES:
Dyspnea Index | 3rd week
  Changes for baseline for level of Shortness of breath is measured using Dyspnea Index. The dyspnea index, also known as the Modified Medical Research Council (MMRC) scale, measures the severity of breathlessness or dyspnea. It's a 5-point scale: Grade 0: No dyspnea, Grade 1: Dyspnea during strenuous exercise, Grade 2: Dyspnea during moderate exercise, Grade 3: Dyspnea during light exercise or walking on level ground, Grade 4: Dyspnea during daily activities or at rest. This scale helps assess the impact of treatment on copd patients.
Tampa Scale of Kinesiophobia | 3rd week
  Changes from baseline for level of kinesiophobia is measured using Tampa scale. The most widely used scale for assessing kinesiophobia is the Tampa Scale of Kinesiophobia (TSK). This questionnaire contains 17 items that gauge a person's fear of movement and associated with movement. Each item is rated on a 4-point Likert scale, with a higher score indicating a greater degree of kinesiophobia. It has an excellent reliability of Cronbach Alpha > 0.9 (18).
  Scores for each item are added together to get a total score. Scores can range from 17 (low kinesiophobia) to 68 (high kinesiophobia). A cut-off score of 37 is often used to indicate high kinesiophobia in COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan institute of medical sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muhammed A, Moiz JA, Singla D, Ali MS, Talwar D. Postural abnormalities in phenotypes of chronic obstructive pulmonary disease. Braz J Phys Ther. 2020 Jul-Aug;24(4):325-332. doi: 10.1016/j.bjpt.2019.05.002. Epub 2019 May 24. PMID 31151892
- [Background] Corlateanu A, Mendez Y, Wang Y, Garnica RJA, Botnaru V, Siafakas N. "Chronic obstructive pulmonary disease and phenotypes: a state-of-the-art.". Pulmonology. 2020 Mar-Apr;26(2):95-100. doi: 10.1016/j.pulmoe.2019.10.006. Epub 2019 Nov 15. PMID 31740261
- [Background] Agusti A, Vogelmeier C, Faner R. COPD 2020: changes and challenges. Am J Physiol Lung Cell Mol Physiol. 2020 Nov 1;319(5):L879-L883. doi: 10.1152/ajplung.00429.2020. Epub 2020 Sep 23. No abstract available. PMID 32964724
- [Background] Brandsma CA, de Vries M, Costa R, Woldhuis RR, Konigshoff M, Timens W. Lung ageing and COPD: is there a role for ageing in abnormal tissue repair? Eur Respir Rev. 2017 Dec 6;26(146):170073. doi: 10.1183/16000617.0073-2017. Print 2017 Dec 31. PMID 29212834
- [Background] Cardoso DM, Fregonezi GA, Jost RT, Gass R, Alberton CL, Albuquerque IM, Paiva DN, Barreto SS. Acute effects of Expiratory Positive Airway Pressure (EPAP) on different levels in ventilation and electrical activity of sternocleidomastoid and parasternal muscles in Chronic Obstructive Pulmonary Disease (COPD) patients: a randomized controlled trial. Braz J Phys Ther. 2016 Nov-Dec;20(6):525-534. doi: 10.1590/bjpt-rbf.2014.0190. Epub 2016 Sep 16. PMID 27683840
- [Background] Shiraishi M, Higashimoto Y, Sugiya R, Mizusawa H, Takeda Y, Fujita S, Nishiyama O, Kudo S, Kimura T, Fukuda K, Tohda Y. Sternocleidomastoid Muscle Thickness Correlates with Exercise Tolerance in Patients with COPD. Respiration. 2023;102(1):64-73. doi: 10.1159/000527100. Epub 2022 Nov 22. PMID 36412608
- [Background] Ahmadipoor A, Khademi-Kalantari K, Rezasoltani A, Naimi SS, Akbarzadeh-Baghban A. Assessing the Reliability of Echo Intensity of Craniovertebral Muscle Group using B-Mode Ultrasound: A Technical Note. J Biomed Phys Eng. 2021 Apr 1;11(2):257-262. doi: 10.31661/jbpe.v0i0.2009-1182. eCollection 2021 Apr. PMID 33937131
- [Background] Tanaka T, Okita M, Jenkins S, Kozu R. Clinical and Psychological Impact of Chronic Pain in People with Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2022 Apr 22;17:893-903. doi: 10.2147/COPD.S359223. eCollection 2022. PMID 35497375
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] Rosa DP, Borstad JD, Pires ED, Camargo PR. Reliability of measuring pectoralis minor muscle resting length in subjects with and without signs of shoulder impingement. Braz J Phys Ther. 2016 Mar 15;20(2):176-83. doi: 10.1590/bjpt-rbf.2014.0146. PMID 26982455